CLINICAL TRIAL: NCT07371403
Title: MB-CART19.1 in Patients With Relapsed/Refractory CD19-positive B Cell Acute Lymphoblastic Leukemia: A Feasibility Study
Brief Title: MB-CART19.1 in Relapsed/Refractory Acute Lymphoblastic Leukemia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Hussein Cancer Center (Other)
Responsible Party: Principal Investigator, Zaid Abdel Rahman, MD, Consultant Hematology, Stem Cell Transplantation and Cellular Therapies, King Hussein Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25KHCC164
Record Dates: First submitted 2026-01-11; First posted 2026-01-27 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Lymphoblastic Leukemia Recurrent; Acute Lymphoblastic Leukemia Refractory; Acute Lymphoblastic Leukemia Not Having Achieved Remission; Acute Lymphoblastic Leukemia With Failed Remission
Keywords: CAR-T; MB-CART19.1; ALL; acute lymphoblastic leukemia; relapsed acute lymphoblastic leukemia; refractory acute lymphoblastic leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MB-CART19.1 (Experimental)
  Interventions: Genetic: MB-CART19.1

INTERVENTIONS:
Genetic: MB-CART19.1 — All participants will undergo leukapheresis for collection of autologous T cells, which will then be manufactured into MB-CART19.1 on-site using CliniMACS Prodigy platform. Successfully manufactured MB-CART19.1 products will be infused back to the patient following a lymphodepleting chemotherapy regimen.

SUMMARY:
Single-arm, prospective, open-label feasibility study evaluating the technical and operational feasibility of manufacturing autologous CD19-directed CAR-T cells (MB-CART19.1) at the point of care for the treatment of relapsed or refractory B-ALL in pediatric and adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 1 year as long as if deemed fit by treating investigator
* CD19 expression must be detected (≥20%) on the malignant cells by flow cytometry.
* Patients with relapsed or refractory disease with >5% blasts in the bone marrow after at least one frontline and one salvage chemotherapy regimen. For patients with Philadelphia-positive disease, a second generation or higher TKI must have been utilized in one of the treatment lines.
* Patients who have relapsed post alloSCT at least 100 days post-transplant, with no evidence of active graft vs host disease, and no longer taking immunosuppressive agents for at least 30 days prior to enrollment.
* Estimated life expectancy > 12 weeks
* Karnofsky or Lansky (age dependent) performance score ≥ 60
* Patients and/or parents must give their written informed consent/assent.
* CNS and/or testicular involvement are allowed, only if cleared and in the presence of systemic involvement.

Exclusion Criteria:

* Rapidly progressive, uncontrolled disease as assessed by the treating physician and/or principal investigator.
* Persistent extramedullary disease.
* Isolated CNS and/or testicular disease.
* Current autoimmune disease, or history of autoimmune disease with potential CNS involvement
* Active hepatitis B, C or HIV
* Active clinically significant CNS dysfunction (including but not limited to uncontrolled seizure disorders, cerebrovascular ischemia or hemorrhage, dementia, paralysis)
* History of an additional malignancy (≤ 3 years) other than non-melanoma skin cancer or carcinoma in situ.
* Pulmonary function: Patients with pre-existing severe lung disease (FEV1 or FVC < 65%) or an oxygen requirement of >28% O2 FiO2 or active pulmonary infection.
* Cardiac function: Left ventricular ejection fraction <50% by echocardiography
* Renal function: Creatinine clearance <50 mL/min/1.73 m2
* Liver function: patients with serum bilirubin ≥3 times upper limit of or AST or ALT > 5 times upper limit of normal, unless due to leukemic liver infiltration as determined by the investigators.
* Pregnant or breast-feeding females
* Medications: systemic chemotherapies, corticosteroids with the exception of physiologic replacement dosing (<0.5 mg/kg/day of methylprednicone), tyrosine kinase inhibitors (TKI) within 7 days prior to leukapheresis, Fludarabine/clofarabine or immunosuppressive drugs and antibodies (e.g. rituximab, blinatumomab) or investigational drugs or donor lymphocyte

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of enrolled patients for whom MB-CART19.1 product is successfully manufactured on-site and meets release criteria. | From patient enrollment through completion of manufacturing and release testing; estimated 2-4 weeks per patient and up to 12 months for the full cohort.
  Assessment of the feasibility and success rate of on-site manufacturing of MB-CART19.1, defined as the proportion of enrolled patients whose cell product is produced and meets established release specifications.

SECONDARY OUTCOMES:
Overall response rate (ORR) (CR, CR with incomplete hematologic recovery (CRh)) on day 28. | Up to approximately 28 days after the last patient infusion.
  Evaluation of overall response rate (ORR) at Day 28, measured as the percentage of patients who achieve complete remission (CR) or complete remission with incomplete hematologic recovery (CRh) following MB-CART19.1 infusion.
Duration of response time from first documented response to progression or death up to 12 months post-infusion | Up to 12 months post-infusion
  Duration of response time from first documented response to progression or death up to 12 months post-infusion
Rate of measurable residual disease (MRD) negativity at 1-, 3-, 6- and 12-month intervals | at 1-, 3-, 6- and 12-month intervals
  Evaluation of rate of measurable residual disease (MRD) negativity at scheduled follow-up visits to monitor clinical status and response post-infusion.
MB-CART19.1 manufacturing turnaround time | From leukapheresis to product release (estimated 2 weeks per patient).
  Time required to complete on-site manufacturing of MB-CART19.1 from leukapheresis to product release.
Overall incidence and severity of adverse events | From infusion through 12 months post-infusion per patient.
  Assessment of the overall incidence and severity of adverse events (AEs) in patients receiving MB-CART19.1, including all treatment-related and non-treatment-related events, graded according to standard toxicity criteria.
Overall incidence and severity of MB-CART19.1- specific adverse events (cytokine release syndrome (CRS)) | From infusion through 12 months post-infusion per patient.
  Assessment of the overall incidence and severity of cytokine release syndrome (CRS) in patients receiving MB-CART19.1, graded according to the American Society for Transplantation and Cellular Therapy (ASTCT) consensus criteria.
Overall incidence and severity MB-CART19.1-specific adverse events (Immune effector cell associated neurotoxicity syndrome (ICANS)) | From infusion through 12 months post-infusion per patient.
  Assessment of the overall incidence and severity of Immune effector cell associated neurotoxicity syndrome (ICANS) in patients receiving MB-CART19.1, graded according to the American Society for Transplantation and Cellular Therapy (ASTCT) consensus criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Zaid Abdel Rahman, Consultant,Hematology/Oncology, Principal Investigator — King Hussein Cancer Center; Dr. Hasan Hashem, Consultant,Hematology/Oncology, Principal Investigator — King Hussein Cancer Center
Locations (1):
- King Hussein Cancer Center, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided